CLINICAL TRIAL: NCT05376995
Title: Effect of Graston Technique Versus Muscle Energy Technique on Improving Hamstring Flexibility and ADLS in Knee Osteoarthritis
Brief Title: Effect of Graston Technique Versus MET on Improving Hamstring Flexibility and ADLS in Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DPT/Batch-Fall17/511
Record Dates: First submitted 2022-04-24; First posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Comparison of Graston technique versus muscle energy technique among patient of knee osteoarthritis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Graston technique. (Experimental): The Graston Technique is a form of manual therapy known as soft-tissue instrument-assisted mobilization
  Interventions: Diagnostic Test: Graston technique
- muscle energy technique (Experimental): Muscle Energy Technique (MET), uses a muscle's own energy in the form of gentle isometric contractions to relax the muscles via autogenic or reciprocal inhibition and lengthen the muscle
  Interventions: Diagnostic Test: muscle energy technique

INTERVENTIONS:
Diagnostic Test: Graston technique — Graston technique among patient of knee osteoarthritis
  Arms: Graston technique.
Diagnostic Test: muscle energy technique — muscle energy technique among patient of knee osteoarthritis
  Arms: muscle energy technique

SUMMARY:
The objective of this study is to determine the comparison of Graston technique versus muscle energy technique to improve hamstring flexibility and ADL among patient of knee O.A.

ELIGIBILITY:
Inclusion Criteria:

* Knee osteoarthritis patient with bilateral (but tested only severe side) or unilateral limb involvement.(13)
* Knee osteoarthritis patient already diagnosed by orthopedic surgeon with x ray findings showing grade I or II in kellgren and Lawrence criteria for knee OA will be selected. (16)
* Ambulate independently with or without assistive devices and ascend and descend at least a flight of stairs.(13)
* Both male and female will be included in study.
* Age above 40 to 55years.(13)

Exclusion Criteria:

* Patient with history of any known neurological, cardio or respiratory conditions.
* Patient present with history of open wound, Skin infection or tumors in the area of treatment.
* Any other orthopedic condition or fracture in the area of treatment limb.
* Patient will be excluded if they have low back pain, sciatica or deformities related to his spine and knee.
* Patient with history of recent lower limb or spinal surgeries.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
knee osteoarthritis | 6 Months
  Comparison of Graston technique versus muscle energy technique among patient of knee osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaudary Muhammad Akram Teaching Hospital, Lahore, Punjab Province, Pakistan